CLINICAL TRIAL: NCT05340686
Title: Braining - A Randomized Controlled Study on Moderate-vigorous Aerobic Physical Exercise (PE) as an add-on Treatment in Bipolar Disorder. Effects on Recovery Time and Long-term Prevention From Bipolar Depression
Brief Title: Braining- Aerobic Physical Activity as Add on Treatment in Bipolar Depression
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties recruiting
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Braining Bipolar RCT
Record Dates: First submitted 2022-03-31; First posted 2022-04-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder; Bipolar Affective Disorder; Remission in; Bipolar Affective Disorder, Currently Depressed, Moderate
Keywords: physical exercise; physical activity
MeSH Terms: conditions — Bipolar Disorder; Lymphoma, Follicular; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Braining high intensity (Experimental): Moderate to vigorous physical exercise, supervised by psychiatric staff 3 times per week
  Interventions: Behavioral: Aerobic Physical Exercise
- Braining relaxing exercise (Active Comparator): Relaxation, light yoga or stretching exercise, supervised by psychiatric staff 3 times per week
  Interventions: Behavioral: Relaxing Physical Exercise
- Information about physical exercise (Active Comparator): Written and oral information about health benefits from physical exercise, provided by researcher on one occasion.
  Interventions: Behavioral: Information about physical exercise

INTERVENTIONS:
Behavioral: Aerobic Physical Exercise — Moderate to vigorous physical exercise 30-45 minutes in a group setting led by psychiatric staff, 3 times per week for 6 weeks
  Arms: Braining high intensity
Behavioral: Relaxing Physical Exercise — Relaxing exercises (stretching, light yoga) 30-45 minutes in a group setting led by psychiatric staff, 3 times per week for 6 weeks
  Arms: Braining relaxing exercise
Behavioral: Information about physical exercise — Written and oral information about physical exercise recommendations, on one occasion, by researcher
  Arms: Information about physical exercise

SUMMARY:
Hypothesis: the hypothesis of the study is that aerobic physical exercise (PE) performed with the method Braining accelerates recovery from bipolar depression as well as improves psychiatric and somatic health in individuals with bipolar depression Method: a randomized controlled trial with 54 patients with bipolar depression are randomized to 6 weeks of either 1) supervised aerobic PE 3 times/week, 2) supervised relaxation/stretching 3 times/week or 3) information about PE but no supervised activity.

DETAILED DESCRIPTION:
The hypothesis of this study is that adding aerobic PE might accelerate recovery, reduce negative side effects, improve mental wellbeing and function, increase long term prevention against relapsing bipolar episodes and reduce risk for complications such as cardiovascular disease in patients with bipolar disorder. Furthermore the study aims to evaluate if the effect of PE is linked to biological factors such as genetical factors, stress hormone levels, level of inflammation and other biological markers for health and disease that can be measured in standard blood samples.

Patients diagnosed with bipolar disorder with ongoing depression are invited to participate in the study at regular visits in the psychiatric clinic. All study participants are medicated with mood stabilizers according to routine treatment and receive regular treatment for bipolar depression. After informed consent the study participants will be randomized to one of three groups 1) moderate to vigorous PE group training together with psychiatric staff three times per week 2) relaxing and stretching exercises group training together with psychiatric staff three times per week 3) information about PE and relaxation but no supervised PE or relaxation/stretching, for the 6 weeks of the study period.

BEFORE: The first week consists of pre-test including interview regarding medical history and physical and psychiatric examination, ECG and blood samples. To measure level of physical activity the participants wear an activity monitor, Actiheart, that continuously registers physical activity for 7 days. The study participants will also fill out different questionnaires regarding general health and psychiatric symptoms.

STUDY PERIOD: During the 6 weeks long study period the participants fill out an activity questionnaire and health questionnaires once a week.

AFTER: during the sixth week of the study period evaluation is being performed with repetition of the physical and psychiatric examination, blood samples and questionnaires. After 1, 2 and 3 years after the exercise period the questionnaires are repeated. Blood samples are repeated one year after the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Psychiatry Southwest, Karolinska University Hospital Region Stockholm Sweden.
* Bipolar disorder
* Ongoing depression, defined as a PHQ-9 score of 9 or higher at any occasion 2 weeks before inclusion.

Exclusion Criteria:

* Severe psychiatric disorder such as mania and psychosis
* Medical conditions such as heart- and lung diseases where PE is contraindicated.
* Unable to understand written and spoken Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-04-20 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 (Patient Health Questionnaire - 9 items) | Change from inclusion to follow up 6 weeks after inclusion
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.
PHQ-9 (Patient Health Questionnaire - 9 items) | At follow up 12 months after intervention.
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.
PHQ-9 (Patient Health Questionnaire - 9 items) | At follow up 24 months after intervention.
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.
PHQ-9 (Patient Health Questionnaire - 9 items) | At follow up 36 months after intervention.
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.

SECONDARY OUTCOMES:
MADRS (Montgomery-Åsberg Depression Rating Scale) | Change from inclusion to follow up 6 weeks after inclusion
  Clinician-rated scale to assess degree of depressive symptoms. 10 items. Minimum value 0 and maximum value 60, where higher values indicate more depressive symptoms.
AS-18 (Affective self rating scale) | Change from inclusion to follow up 6 weeks after inclusion
  Self-assessment of symptoms of depression and hypomania/mania. 9 items for depression and 9 items for mania. Score 0-72. A score of over 10 on the depressive or manic/hypomanic subscale should give rise to suspicion of ongoing depression and hypomania/mania respectively. Scores of over 10 on both the depressive and manic/hypomanic scale at the same time give may indicate an affective mixed state.
AS-18 (Affective self rating scale) | At follow up 12 months after intervention.
  Self-assessment of symptoms of depression and hypomania/mania. 9 items for depression and 9 items for mania. Score 0-72. A score of over 10 on the depressive or manic/hypomanic subscale should give rise to suspicion of ongoing depression and hypomania/mania respectively. Scores of over 10 on both the depressive and manic/hypomanic scale at the same time give may indicate an affective mixed state.
AS-18 (Affective self rating scale) | At follow up 24 months after intervention.
  Self-assessment of symptoms of depression and hypomania/mania. 9 items for depression and 9 items for mania. Score 0-72. A score of over 10 on the depressive or manic/hypomanic subscale should give rise to suspicion of ongoing depression and hypomania/mania respectively. Scores of over 10 on both the depressive and manic/hypomanic scale at the same time give may indicate an affective mixed state.
AS-18 (Affective self rating scale) | At follow up 36 months after intervention.
  Self-assessment of symptoms of depression and hypomania/mania. 9 items for depression and 9 items for mania. Score 0-72. A score of over 10 on the depressive or manic/hypomanic subscale should give rise to suspicion of ongoing depression and hypomania/mania respectively. Scores of over 10 on both the depressive and manic/hypomanic scale at the same time give may indicate an affective mixed state.
YMRS (Young Ziegler Mania Rating Scale) | Change from inclusion to follow up 6 weeks after inclusion
  Interviewer-rated scale. Includes 11 items; seven are rated from 0 (absent) to 4; four from 0 to 8; total scores range from 0 to 60. A higher value indicates worse symptoms of hypomania/mania.
YMRS (Young Ziegler Mania Rating Scale) | At follow up 12 months after intervention.
  Interviewer-rated scale. Includes 11 items; seven are rated from 0 (absent) to 4; four from 0 to 8; total scores range from 0 to 60. A higher value indicates worse symptoms of hypomania/mania.
YMRS (Young Ziegler Mania Rating Scale) | At follow up 24 months after intervention.
  Interviewer-rated scale. Includes 11 items; seven are rated from 0 (absent) to 4; four from 0 to 8; total scores range from 0 to 60. A higher value indicates worse symptoms of hypomania/mania.
YMRS (Young Ziegler Mania Rating Scale) | At follow up 36 months after intervention.
  Interviewer-rated scale. Includes 11 items; seven are rated from 0 (absent) to 4; four from 0 to 8; total scores range from 0 to 60. A higher value indicates worse symptoms of hypomania/mania.
CGI-S (Clinical Global Impressions - Severity Scale) | Change from inclusion to follow up 6 weeks after inclusion
  A one-item clinician assessed measure which evaluates the severity of psychopathology from 1 to 7, where 1 is 'normal' and 7 is 'among the most extremely ill patients' by the question "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?".
CGI-S (Clinical Global Impressions - Severity Scale) | At follow up 12 months after intervention
  A one-item clinician assessed measure which evaluates the severity of psychopathology from 1 to 7, where 1 is 'normal' and 7 is 'among the most extremely ill patients' by the question "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?".
CGI-S (Clinical Global Impressions - Severity Scale) | At follow up 24 months after intervention
  A one-item clinician assessed measure which evaluates the severity of psychopathology from 1 to 7, where 1 is 'normal' and 7 is 'among the most extremely ill patients' by the question "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?".
CGI-S (Clinical Global Impressions - Severity Scale) | At follow up 36 months after intervention
  A one-item clinician assessed measure which evaluates the severity of psychopathology from 1 to 7, where 1 is 'normal' and 7 is 'among the most extremely ill patients' by the question "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?".
Blood pressure | Change from inclusion to follow up 6 weeks after inclusion
  systolic and diastolic, mmHg
Blood pressure | At follow up 12 months after intervention
  systolic and diastolic, mmHg
Blood pressure | At follow up 24 months after intervention
  systolic and diastolic, mmHg
Blood pressure | At follow up 36 months after intervention
  systolic and diastolic, mmHg
Heart rate | Change from inclusion to follow up 6 weeks after inclusion
  Heart rate, beats per minute
Heart rate | At follow up 12 months after intervention
  Heart rate, beats per minute
Heart rate | At follow up 24 months after intervention
  Heart rate, beats per minute
Heart rate | At follow up 36 months after intervention
  Heart rate, beats per minute
BMI (Body mass index) | Change from inclusion to follow up 6 weeks after inclusion
  Weight in kg divided by the square of height in m
BMI (Body mass index) | At follow up 12 months after intervention
  Weight in kg divided by the square of height in m
BMI (Body mass index) | At follow up 24 months after intervention
  Weight in kg divided by the square of height in m
BMI (Body mass index) | At follow up 36 months after intervention
  Weight in kg divided by the square of height in m
Waist circumference | Change from inclusion to follow up 6 weeks after inclusion
  Waist circumference, cm
Waist circumference | At follow up 12 months after intervention
  Waist circumference, cm
Waist circumference | At follow up 24 months after intervention
  Waist circumference, cm
Waist circumference | At follow up 36 months after intervention
  Waist circumference, cm
FBS (fasting blood sugar) | Change from inclusion to follow up 6 weeks after inclusion
  fasting blood sugar, mmol/l
FBS (fasting blood sugar) | At follow up 12 months after intervention.
  fasting blood sugar, mmol/l
FBS (fasting blood sugar) | At follow up 24 months after intervention.
  fasting blood sugar, mmol/l
FBS (fasting blood sugar) | At follow up 36 months after intervention.
  fasting blood sugar, mmol/l
HbA1c (Hemoglobin A1c) | Change from inclusion to follow up 6 weeks after inclusion
  Glycated hemoglobin, mmol/mol
HbA1c (Hemoglobin A1c) | At follow up 12 months after intervention.
  Glycated hemoglobin, mmol/mol
HbA1c (Hemoglobin A1c) | At follow up 24 months after intervention.
  Glycated hemoglobin, mmol/mol
HbA1c (Hemoglobin A1c) | At follow up 36 months after intervention.
  Glycated hemoglobin, mmol/mol
Blood lipids | Change from inclusion to follow up 6 weeks after inclusion
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
Blood lipids | At follow up 12 months after intervention.
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
Blood lipids | At follow up 24 months after intervention.
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
Blood lipids | At follow up 36 months after intervention.
  Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, mmol/L
CRP (C-reactive protein) | Change from inclusion to follow up 6 weeks after inclusion
  Measurement of inflammation and infection, mmol/L
CRP (C-reactive protein) | At follow up 12 months after intervention.
  Measurement of inflammation and infection, mmol/L
CRP (C-reactive protein) | At follow up 24 months after intervention.
  Measurement of inflammation and infection, mmol/L
CRP (C-reactive protein) | At follow up 36 months after intervention.
  Measurement of inflammation and infection, mmol/L
Telomere length | Change from inclusion to follow up 6 weeks after inclusion
  telomere length in leukocytes
Telomere length | At follow up 12 months after intervention.
  telomere length in leukocytes
Telomerase | Change from inclusion to follow up 6 weeks after inclusion
  Enzyme activity in blood
Telomerase | At follow up 12 months after intervention.
  Enzyme activity in blood
WHODAS 2.0 (World health organization disability assessment schedule) | Change from inclusion to follow up 6 weeks after inclusion
  Self rated disability. Minimum value 0, maximum value 100, where higher values indicate more disability.
WHODAS 2.0 (World health organization disability assessment schedule) | At follow up 12 months after intervention.
  Self rated disability. Minimum value 0, maximum value 100, where higher values indicate more disability.
WHODAS 2.0 (World health organization disability assessment schedule) | At follow up 24 months after intervention.
  Self rated disability. Minimum value 0, maximum value 100, where higher values indicate more disability.
WHODAS 2.0 (World health organization disability assessment schedule) | At follow up 36 months after intervention.
  Self rated disability. Minimum value 0, maximum value 100, where higher values indicate more disability.
EQ-5D-5L (EuroQol VAS) | Change from inclusion to follow up 6 weeks after inclusion
  Self-assessment instrument for describing and valuing health. Defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Also included is an overall health rating on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 55555 (worst health). A number of methods exist for analysing these five digit profiles. However, frequently they are converted to a single utility index using country specific value sets. A higher index number indicates a poorer self-assessed health.
EQ-5D-5L (EuroQol VAS) | At follow up 12 months after intervention.
  Self-assessment instrument for describing and valuing health. Defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Also included is an overall health rating on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 55555 (worst health). A number of methods exist for analysing these five digit profiles. However, frequently they are converted to a single utility index using country specific value sets. A higher index number indicates a poorer self-assessed health.
EQ-5D-5L (EuroQol VAS) | At follow up 24 months after intervention.
  Self-assessment instrument for describing and valuing health. Defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Also included is an overall health rating on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 55555 (worst health). A number of methods exist for analysing these five digit profiles. However, frequently they are converted to a single utility index using country specific value sets. A higher index number indicates a poorer self-assessed health.
EQ-5D-5L (EuroQol VAS) | At follow up 36 months after intervention.
  Self-assessment instrument for describing and valuing health. Defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Also included is an overall health rating on a 0-100 hash-marked, vertical visual analogue scale (EQ-VAS). Assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 55555 (worst health). A number of methods exist for analysing these five digit profiles. However, frequently they are converted to a single utility index using country specific value sets. A higher index number indicates a poorer self-assessed health.
SRH (Self-rated health) | Change from inclusion to follow up 6 weeks after inclusion
  SRH is typically measured as a single-item, the most common wording of which is "In general, would you say your health is" with the response items "excellent," "very good," "good," "fair," or "poor."
SRH (Self-rated health) | At follow up 12 months after intervention.
  SRH is typically measured as a single-item, the most common wording of which is "In general, would you say your health is" with the response items "excellent," "very good," "good," "fair," or "poor."
SRH (Self-rated health) | At follow up 24 months after intervention.
  SRH is typically measured as a single-item, the most common wording of which is "In general, would you say your health is" with the response items "excellent," "very good," "good," "fair," or "poor."
SRH (Self-rated health) | At follow up 36 months after intervention.
  SRH is typically measured as a single-item, the most common wording of which is "In general, would you say your health is" with the response items "excellent," "very good," "good," "fair," or "poor."
BBQ (Brunnsviken Brief Quality of Life Questionnaire) | Change from inclusion to follow up 6 weeks after inclusion
  Self rated quality of life. Minimum value 0, maximum value 96, where higher values indicate higher quality of life satisfaction.
BBQ (Brunnsviken Brief Quality of Life Questionnaire) | At follow up 12 months after intervention.
  Self rated quality of life. Minimum value 0, maximum value 96, where higher values indicate higher quality of life satisfaction.
BBQ (Brunnsviken Brief Quality of Life Questionnaire) | At follow up 24 months after intervention.
  Self rated quality of life. Minimum value 0, maximum value 96, where higher values indicate higher quality of life satisfaction.
BBQ (Brunnsviken Brief Quality of Life Questionnaire) | At follow up 36 months after intervention.
  Self rated quality of life. Minimum value 0, maximum value 96, where higher values indicate higher quality of life satisfaction.
Occupational level measured in % of work ability in medical certificate | Change from inclusion to follow up 6 weeks after inclusion
  Complete sick leave 0%, partial sick leave 25-75 %, completely able to work 100%.
Occupational level measured in % of work ability in medical certificate | At follow up 12 months after intervention.
  Complete sick leave 0%, partial sick leave 25-75 %, completely able to work 100%.
Occupational level measured in % of work ability in medical certificate | At follow up 24 months after intervention.
  Complete sick leave 0%, partial sick leave 25-75 %, completely able to work 100%.
Occupational level measured in % of work ability in medical certificate | At follow up 36 months after intervention.
  Complete sick leave 0%, partial sick leave 25-75 %, completely able to work 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Martinsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Region Stockholm, Psykiatri Sydväst (Psychiatric Clinic Psychiatry Southwest), Stockholm, Stockholm County, Sweden